CLINICAL TRIAL: NCT06832878
Title: Postoperative Oral Tranexamic Acid in Patients Undergoing Primary Total Joint Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joshua S. Bingham, Associate Professor of Orthopedics, Orthopedic Consultant, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-008865
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Arthroplasty
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral tranexamic acid (Experimental)
  Interventions: Drug: Oral Tranexamic Acid
- Control Group (No Intervention)

INTERVENTIONS:
Drug: Oral Tranexamic Acid — Subjects will receive a 1.95 g dose of oral TXA at the following timepoints: (1) following ambulation, (2) postoperative day 1, (3) postoperative day 2, and (4) postoperative day 3
  Arms: Oral tranexamic acid

SUMMARY:
The purpose of this study is to evaluate the impact of an extended oral Tranexamic Acid regimen on patient reported outcome scores, time to independent ambulation, postoperative range of motion, swelling, change in hemoglobin levels, 90-day complications, readmission and reoperation.

ELIGIBILITY:
Inclusion Criteria

* Adults aged > 18 years (All women of childbearing potential undergo pregnancy testing prior to THA as per our institutional protocol)
* Written informed consent
* Patients undergoing primary THA diagnosis of end-stage osteoarthritis
* Patients receiving spinal anesthesia
* Patients being discharged on postoperative day 1

Exclusion Criteria

* Patients with a TXA allergy
* Patients undergoing revision procedures
* Patients undergoing primary THA for a diagnosis other than end-stage osteoarthritis
* Patients receiving general anesthesia
* Patients being discharged on the same day of surgery
* Cancer patients
* Patients with a history of prior VTE event
* Patients on preoperative anticoagulants other than ASA
* Pregnant patients (All women of child bearing potential undergo pregnancy testing prior to THA as per our institutional protocol)
* Female patients who are on hormonal contraception
* Patients with history of retinal vein or artery occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score | Baseline, 3 days postoperative, 2 weeks, 6 weeks, 12 weeks
  The VAS is a 11-item questionnaire assessing pain. Using a scale of 0 = no pain to 10 = worst pain. Total scores range from 0 - 110, lower scores indicating lower pain and higher scores indicating greater pain.
Hip Disability and Osteoarthritis Outcome Score (HOOS) for Joint Replacement (JR) | Baseline, 3 days postoperative, 2 weeks, 6 weeks, 12 weeks
  The Hip Disability and Osteoarthritis Outcome Score (HOOS) for Joint Replacement (JR) is a questionnaire designed to measure outcomes for patients with hip replacements. Results are scored 0-11. 0 = total hip disability, 100 = perfect hip health.

SECONDARY OUTCOMES:
Hemoglobin | Baseline, prior to discharge, day 3 postoperatively
  Hemoglobin is a protein within red blood cells. As glucose enters the bloodstream, it binds to hemoglobin, or glycates. The more glucose that enters the bloodstream, the higher the amount of glycated hemoglobin. An A1C level below 5.7 percent is considered normal. Reported as percentage of glycated hemoglobin
Harris Hip Score (HHS) | Baseline, 3 days postoperative, 2 weeks, 6 weeks, 12 weeks
  The Harris Hip Score (HHS) is a tool used to assess hip function and the results of hip treatments, such as hip replacements. It's a 100-point scale that measures four areas: pain, function, deformity, and range of motion. A higher score indicates less dysfunction and better outcomes. A score of less than 70 is considered poor, 70-80 is fair, 80-90 is good, and 90-100 is excellent.
Short Form Health Survey (SF-12) | Baseline, 3 days postoperative, 2 weeks, 6 weeks, 12 weeks
  The 12-Item Short Form Health Survey (SF-12) is a questionnaire which consists of 12 questions covering physical and mental health domains. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
Time to Independent Ambulation | 12 weeks
  Duration of time post-operation until the subject can walk without any support or assistance, reported in days
Oxford Hip Score | Baseline, 3 days postoperative, 2 weeks, 6 weeks, 12 weeks
  The Oxford Hip Score (OHS) is a standard patient-reported outcome (PRO) measure, or PROM, developed to assess function and pain in patients undergoing total hip replacement (THR) surgery, particularly in the context of clinical trials. The OHS has also been used for the assessment of patient outcomes, including physical therapy, and use of joint supplements (disease specific and general health measure are two other outcome measures).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Bingham, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials